CLINICAL TRIAL: NCT01149538
Title: Postnatal Choline Supplementation in Children With Prenatal Alcohol Exposure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0910M73517; R21AA019580 (NIH)
Record Dates: First submitted 2010-06-21; First posted 2010-06-23 (Estimated); Results first posted 2016-08-11 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-10

CONDITIONS: Fetal Alcohol Spectrum Disorders; Fetal Alcohol Syndrome; Partial Fetal Alcohol Syndrome; Alcohol Related Neurodevelopmental Disorder; Prenatal Alcohol Exposure
Keywords: FASD; FAS; Alcohol; Prenatal Alcohol
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders | interventions — Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Choline Bitartrate (Experimental): Choline Bitartrate supplementation
  Interventions: Drug: Choline bitartrate
- Placebo (Placebo Comparator): Placebo for choline bitartrate supplementation
  Interventions: Dietary Supplement: Placebo for choline bitartrate

INTERVENTIONS:
Drug: Choline bitartrate — Choline bitartrate 500 mg. daily, administered in fruit-flavored drink mix.
  Arms: Choline Bitartrate
Dietary Supplement: Placebo for choline bitartrate — Placebo for choline bitartrate, administered daily in fruit-flavored drink mix.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if choline bitartrate can be administered daily to children with prenatal alcohol exposure, ages 2.5 to 5, as a potential treatment for brain development and cognitive functioning.

ELIGIBILITY:
Inclusion Criteria:

* Available parent or legal guardian capable of participating in informed consent process
* Documented history of heavy prenatal alcohol exposure (self-report, social service records, or adoption records) or presence of facial dysmorphology characteristic of FASD or both
* Evidence of cognitive deficit in at least one neurocognitive domain

Exclusion Criteria:

* History of neurological condition (ex. epilepsy, cerebral palsy, traumatic brain injury)
* History of medical condition known to affect brain function
* History of other neurodevelopmental disorder (ex. autism, down syndrome)
* History of very low birthweight (<1500 grams)
* History of prenatal exposure to drugs other than alcohol, nicotine, and caffeine

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Wozniak, Ph.D., Principal Investigator — University of Minnesota; Michael Georgieff, M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Wozniak JR, Eckerle JK, Gimbel BA, Ernst AM, Anthony ME, Tuominen KA, de Water E, Zeisel SH, Georgieff MK. Choline enhances elicited imitation memory performance in preschool children with prenatal alcohol exposure: a cumulative report of 3 randomized controlled trials. Am J Clin Nutr. 2025 Apr;121(4):921-931. doi: 10.1016/j.ajcnut.2025.02.009. Epub 2025 Feb 14. PMID 39956364
- [Derived] Gimbel BA, Anthony ME, Ernst AM, Roediger DJ, de Water E, Eckerle JK, Boys CJ, Radke JP, Mueller BA, Fuglestad AJ, Zeisel SH, Georgieff MK, Wozniak JR. Long-term follow-up of a randomized controlled trial of choline for neurodevelopment in fetal alcohol spectrum disorder: corpus callosum white matter microstructure and neurocognitive outcomes. J Neurodev Disord. 2022 Dec 16;14(1):59. doi: 10.1186/s11689-022-09470-w. PMID 36526961
- [Derived] Smith SM, Virdee MS, Eckerle JK, Sandness KE, Georgieff MK, Boys CJ, Zeisel SH, Wozniak JR. Polymorphisms in SLC44A1 are associated with cognitive improvement in children diagnosed with fetal alcohol spectrum disorder: an exploratory study of oral choline supplementation. Am J Clin Nutr. 2021 Aug 2;114(2):617-627. doi: 10.1093/ajcn/nqab081. PMID 33876196
- [Derived] Wozniak JR, Fink BA, Fuglestad AJ, Eckerle JK, Boys CJ, Sandness KE, Radke JP, Miller NC, Lindgren C, Brearley AM, Zeisel SH, Georgieff MK. Four-year follow-up of a randomized controlled trial of choline for neurodevelopment in fetal alcohol spectrum disorder. J Neurodev Disord. 2020 Mar 12;12(1):9. doi: 10.1186/s11689-020-09312-7. PMID 32164522
- [Derived] Wozniak JR, Fuglestad AJ, Eckerle JK, Fink BA, Hoecker HL, Boys CJ, Radke JP, Kroupina MG, Miller NC, Brearley AM, Zeisel SH, Georgieff MK. Choline supplementation in children with fetal alcohol spectrum disorders: a randomized, double-blind, placebo-controlled trial. Am J Clin Nutr. 2015 Nov;102(5):1113-25. doi: 10.3945/ajcn.114.099168. Epub 2015 Oct 7. PMID 26447156

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Choline Bitartrate | Placebo
Started | 31 | 29
Completed | 26 | 25
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Choline Bitartrate | Placebo | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.79 (.80) | 3.92 (.76) | 3.855 (.78)
Gender [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Side Effects of Choline Bitartrate
Description: Side effects of choline bitartrate will be monitored by the study physician and the P.I. with physical examinations and telephone contact.
Time Frame: Baseline, 6 months, & 9 months
Population: Children with fetal alcohol spectrum disorders receiving either choline or placebo for 9 months
Measure: Number; unit: participants
Arm/Group | Choline Bitartrate | Placebo
Number analyzed (Participants) | 31 | 29
participants
  Baseline energy level problems | 8 | 10
  6 month energy level problems | 8 | 9
  9 months energy level problems | 8 | 9
  Baseline pain | 3 | 4
  6 month pain | 3 | 4
  9 month pain | 3 | 4
  Baseline skin problems | 6 | 6
  6 month skin problems | 6 | 5
  9 month skin problems | 6 | 5
  Baseline Ear Nose Throat problems | 1 | 0
  6 month Ear Nose Throat problems | 1 | 0
  9 month Ear Nose Throat problems | 1 | 1
  Baseline headaches/dizziness | 2 | 2
  6 month headaches/dizziness | 2 | 2
  9 month headaches/dizziness | 2 | 2
  Baseline vision problems | 2 | 2
  6 month vision problems | 0 | 2
  9 month vision problems | 0 | 2
  Baseline cardiovascular | 1 | 1
  6 month cardiovascular | 1 | 1
  9 month cardiovascular | 1 | 1
  Baseline respiratory problems | 6 | 6
  6 month respiratory problems | 6 | 6
  9 month respiratory problems | 6 | 6
  Baseline gastrointestinal problems | 18 | 14
  6 month gastrointestinal problems | 18 | 11
  9 month gastrointestinal problems | 18 | 11
  Baseline genitourinary problems | 4 | 9
  6 month genitourinary problems | 4 | 8
  9 month genitourinary problems | 4 | 8
  Baseline musculoskeletal problems | 0 | 1
  6 month musculoskeletal problems | 0 | 1
  9 month musculoskeletal problems | 0 | 1
  6 month neurologic/psychiatric problems | 11 | 9
  9 month neurologic/psychiatric problems | 11 | 9
  Baseline neurologic/psychiatric problems | 11 | 9
  Baseline allergic problems | 2 | 3
  6 month allergic problems | 0 | 3
  9 month allergic problems | 0 | 3

2. Primary Outcome: Mullen Scales of Early Learning - Early Learning Composite
Description: The Mullen Scales of Early Learning is a measure of global cognitive development and is a primary outcome measure. The Early Learning Composite is the total score for this measure. It is a scaled score with a mean of 100 and a standard deviation of 15 (higher scores indicate better global cognitive status; average range is 85-115; Impaired range is 70 or below; full range is typically 50 - 150, although minimum and maximum scores are dependent on age). See the Mullen Scales reference manual for more psychometric details.
Time Frame: Baseline and 9 months
Population: Including those with partial completion (drop-outs and lost-to-followup).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Choline Bitartrate | Placebo
Number analyzed (Participants) | 31 | 29
units on a scale
  Baseline | 83.2 (13.7) | 84.3 (21.4)
  9-month follow-up | 87.1 (16.4) | 89.6 (21.6)

3. Secondary Outcome: Elicited Imitation Task Memory
Description: The Elicited Imitation (EI) paradigm (P.J. Bauer, 1989, Dev. Psychology) was used to measure memory in the participants at baseline, 6 months, and 9 months. The measures were items recalled after a delay (delayed items) and pairs of items recalled after a delay (delayed pairs). The sample was split by age in the analysis (young vs. old) as reflected in the outcome data. Outcome data measures included here are the slopes of the regression lines reflecting change over the three timepoints, controlling for immediate memory performance on the EI task.The slopes are given, as opposed to the raw scores, because these were the values used in the growth curve analyses. Details of these analyses are included in Wozniak et al. (2015) AJCN, doi:10.3945/ajcn.114.099168. NOTE that the means presented below represent the simple slopes that estimate the change in task performance (% of items correct) per 6-month unit of time. To estimate change in task performance over 9 months, multiply by 1.5.
Time Frame: Baseline, 6 months, and 9 months
Population: Young choline group (n=17); Young placebo group (n=13); Old choline group (n=14); Old placebo group (n=16).
Measure: Mean (Standard Error); unit: Slope
Arm/Group | Choline Bitartrate | Placebo
Number analyzed (Participants) | 31 | 29
Slope
  Delayed-Items-Young | 14.24 (3.84) | 4.43 (4.04)
  Delayed-Items-Old | -.71 (3.98) | 4.23 (3.90)
  Delayed-Pairs-Young | 18.97 (3.65) | 10.39 (4.00)
  Delayed-Pairs-Old | 2.69 (3.79) | 7.79 (3.73)
  Immed-Items-Young | 8.48 (4.23) | 13.72 (4.41)
  Immed-Items-Old | 2.59 (4.36) | 3.89 (4.24)
  Immed-Pairs-Young | 8.75 (4.45) | 20.01 (4.80)
  Immed-Pairs-Old | 11.46 (4.61) | 5.50 (4.46)

4. Secondary Outcome: Evoked Response Potentials Microvolts
Description: Evoked response potentials were measured for the memory task. Frontal positive slow-wave potential negative component amplitude data are included.
Time Frame: Baseline, 6 months, and 9 months
Population: Children with FASD who were administered Evoked Response Potential test and provided usable date (choline and placebo arms)
Measure: Mean (Standard Deviation); unit: Mircovolts
Arm/Group | Choline Bitartrate | Placebo
Number analyzed (Participants) | 36 | 35
Mircovolts
  Frontal Positive Slow Wave (PSW) - Baseline | -2.05 (5.49) | 0.57 (7.24)
  Frontal Positive Slow Wave (PSW) - 6 months | -1.04 (4.58) | -1.03 (3.48)
  Frontal Positive Slow Wave (PSW) - 9 months | -0.26 (5.01) | -1.41 (5.23)
  Frontal Neg Component Amplitude - Baseline | -2.53 (5.66) | 0.62 (7.56)
  Frontal Neg Component Amplitude - 6 months | 1.22 (5.46) | -0.84 (4.94)
  Frontal Neg Component Amplitude - 9 months | 0.35 (5.53) | -1.37 (5.08)

5. Secondary Outcome: Evoked Response Potential - Negative Component Latency
Description: Evoked Response Potential - negative component latency data are included.
Time Frame: Baseline, 6 months, and 9 months
Population: Children with FASD who were administered Evoked Response Potential test and provided usable data (choline and placebo arms)
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Choline Bitartrate | Placebo
Number analyzed (Participants) | 36 | 35
Milliseconds
  Frontal Neg Component Latency at baseline | 2.23 (43.96) | 5.35 (60.21)
  Frontal Neg Component at 6 months | 32.45 (60.31) | -4.28 (55.22)
  Frontal Neg Component at 9 months | -4.00 (42.30) | -3.03 (79.62)

ADVERSE EVENTS:
Time Frame: Adverse events reported here represent events EVER reported over the 9-month duration of the study.
Description: Adverse events by organ system (percentage EVER reporting symptoms within each organ system listed - over 9 months). Events were collected in categories listed below (some include multiple symptoms). Individual symptom data exists in detailed notes for each participant but is not available in tallied form (except as aggregated into categories).
Arm/Group | Choline Bitartrate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 15/31 | 13/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Choline Bitartrate (N=31) | Placebo (N=29)
Skip problems (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) — Rash, sweating, nail changes
Ear (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Sore throat, congestion, eye watering, dry eyes
Cardiovascular (Cardiac disorders) | 1 (1) | 0 (0) — Heart racing, rhythm disturbance, swelling
Respiratory (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) — Shortness of breath, wheezing, cough
Gastrointestinal (Gastrointestinal disorders) | 9 (9) | 7 (7) — upset stomach, salivary changes, appetite change, diarrhea, constipation
Fishy Body Odor (Gastrointestinal disorders) | 15 (15) | 1 (1) — Fishy body odor (a common result of choline supplementation)
Genitourinary (Renal and urinary disorders) | 3 (3) | 8 (8) — changes in urination pattern, incontinence, color changes
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) — pain, joint swelling, weakness, cramps
Neurologic (Nervous system disorders) | 6 (6) | 4 (4) — seizures, coordination problems, worsening of mood/behavior
Allergy (Immune system disorders) | 0 (0) | 2 (2) — flushing, itching, changes in tolerance to heat or cold

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No